CLINICAL TRIAL: NCT04479371
Title: Prospective Randomized Trial of Penile Nerve Block With Liposomal Bupivacaine for Hypospadias Repair vs Standard Penile Block With Bupivacaine
Brief Title: Liposomal Bupivacaine vs Standard Penile Block for Hypospadias Repair
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Limited funding and resources to complete FDA requirements for enrollment
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Craig Peters, Chief of Pediatric Urology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU-2020-0686
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Two arms with one receiving liposomal bupivacaine in their penile block vs one receiving standard bupivacaine
Who Masked: Participant
Masking Description: Participants will be blinded as to which block they received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal bupivacaine (Experimental): a penile block administered with novel liposomal bupivacaine during hypospadias repair
  Interventions: Drug: Liposomal bupivacaine
- Standard Penile Block (Active Comparator): Standard weight based bupivacaine penile block during hypospadias repair
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Injecting liposomal bupivacaine for a penile block for analgesia for hypospadias repair
  Other Names: exparel
  Arms: Liposomal bupivacaine
Drug: Bupivacaine — Standard bupivacaine
  Other Names: 0.25% Bupivacaine
  Arms: Standard Penile Block

SUMMARY:
The investigator proposes a prospective randomized study of males with hypospadias to either bupivacaine penile block or liposomal bupivacaine block for hypospadias repair, Figure 3. The investigator will use an envelope system for randomizing 1:1 to either group.

Approach to surgery will be determined by the location of the urethral meatus and degree of chordee along with the amount of skin available and provider preference. Patients who have an ASA classification of 3 or greater, renal or hepatic dysfunction, less than 6 months of age, or refuse the risk of using liposomal bupivacaine during the procedure will be excluded.

The goal is to compare the pain scores of standard bupivacaine penile blocks versus liposomal bupivacaine penile blocks for patients undergoing hypospadias surgery. This is also an opportunity to use liposomal bupivacaine in children as a regional local block for penile surgery. Patients will be enrolled at Children's Medical Center from July 1st, 2019 until 100 total patients are accrued, as specified in our sample size calculation. It is estimated that the trial will be completed in five years with hopes of potentially reaching 100 patients within two years.

DETAILED DESCRIPTION:
Male patients who are greater than 6 months of age will be enrolled in the study prior to elective outpatient hypospadias repair with ASA class 1-2. For a male who meets the inclusion criteria, after informed consent is obtained, he will be randomized at a 1:1 basis to standard penile block with bupivacaine or penile block with liposomal bupivacaine. All patients will be pre-medicated per standard practice with 0.1-0.2 mg PO hydrocodone and 0.25-0.35 mg PO versed.

* Control patients will receive a standardized amount of 0.25% bupivacaine based on age-based ideal body weight calculated as follows: 6 months to 1 year old, 2.5 mg/kg; >1-year-old, 3 mg/kg. Calculating volume of agent that can be administered in mL = allowable ideal body weight dose (mg/kg) x (weight in kg) x (1/ concentration of local anesthetic agent). For example, the average 9-month old male is around 9 kg, therefore, they will receive 9 mL of 0.25% bupivacaine (2.5 mg/mL).
* Treatment patients will receive Liposomal Bupivacaine (Exparel) 1.3% (266mg/20mL or 133mg/10mL) based on current PK studies for the agent. A dose of 4mg/kg will be used. For example, using the fact that the average 9-month old is around 9kg the patient would receive 2.7 mL of liposomal bupivacaine. Since the liposomal bupivacaine has a delayed onset of action, the patients in this arm would receive 0.25% bupivacaine for the immediate analgesic needed for the operative procedure. According to the prescribing information for Pacira pharmaceuticals, bupivacaine HCl can be administered immediately before or in the same syringe as liposomal bupivacaine (Exparel). This is only true as long as the ratio of bupivacaine HCl to Liposomal bupivacaine (Experal) dose does not exceed 1:2 ratio of the agents. Also, a 10mL vial of liposomal bupivacaine (Experal) contains 133mg of free base bupivacaine, which is the molar equivalent of 150mg of bupivacaine HCl. (reference Pacira prescribing information) Therefore, if the dose of 2.7ml of liposomal bupivacaine is used for a 9kg child, then the patient is allowed up to 18mg of bupivacaine HCl to be mixed with the liposomal bupivacaine (1:2 ration or 50% rule from Pacira prescribing information). Our patients will receive a 0.25% bupivacaine dosage that will be calculated using the ideal body weight calculation as stated above, but instead of using 2.5mg/kg dosage it would need to be 2mg/kg so the 50% ratio is met to fit the pharmacodynamics of using liposomal bupivacaine in a safe and predictable manner. Therefore, for the 9kg patient, he would receive 2.7 mL of liposomal bupivacaine and 7.2 mL of 0.25% bupivacaine for a total volume of 9.9 mL of total volume.
* Using the 0.25% bupivacaine in the control arm and experimental arm allows the volume of the local anesthetic to be close in-between the cohorts and ideal for giving a complete penile ring block, since the volume of liposomal bupivacaine needed is very small. The use of 0.25% bupivacaine is important in the liposomal bupivacaine arm, because the liposomal bupivacaine has a delayed release and could not offer local anesthesia until closer to 45 minutes after application. This could potentially lead to patients requiring more systemic anesthesia if liposomal bupivacaine is used alone. Therefore, like many other pediatric providers using liposomal bupivacaine, it will be given in conjunction with 0.25% bupivacaine to improve immediate local anesthesia.
* To standardize the technique of the blocks, each block will be given in the same fashion by each of the pediatric urology providers.

  1. Enrollment and Consenting:
* Patients that fit the inclusion criteria will have the trial discussed with them in the preoperative consultation room with the attending urologist. If the patients' consent to being enrolled, they will receive a copy of the Face, Legs, Activities, Cry, Consolability (FLACC) scale, the post procedure log sheet for the study to record the FLACC scores and PRN medication doses and indication for PRN medication administration, and they will also be shown a video on how to use the FLACC scoring system.
* One of the concerns for using the FLACC as an outcome measure of postoperative pain and a measure of how effective liposomal bupivacaine is in comparison to bupivacaine alone, is the intra-operator differences among patients' parents and reporting a score. We are attempting to control for this by showing a video with an example patient and scoring of this patient for each family to view. This video will be available to enrolled families via email so they can show it to other family members or caregivers (potentially grandparents or nanny/babysitters) who may be scoring the child in the post-operative period, but were not present on the day of surgery, or during the preoperative consultation.

Day of Surgery

* The parent/LAR will most likely be approached for consenting at the preoperative consultation, but will be given ample time to consider, and we will verify they continue to desire to participate on the day of their surgery by the research fellow.
* After the patient is enrolled, the research fellow will pull the next envelope to determine which group each patient will be assigned to.
* The anesthesia team will receive the treatment arm assignment 0.25% bupivacaine HCl alone vs. 0.25% bupivacaine and 1.3% liposomal bupivacaine from the research team member. And enter the order for local anesthetic agent in Epic that will be used during the surgery for the penile block with the appropriate patient weight.
* The agent will be processed by pharmacy and dispensed to the OR for the urologist to administer as a penile ring block at the induction of anesthesia. The urologist and anesthesiologist will be aware of the agent given to the patient for safety concerns, but this should not interfere with trial endpoints since scores will be awarded by the parents who are blinded to the anesthetic agent used.
* The block will be administered in a standard fashion (ring block) by the pediatric urologist in either arm of the study.

  2. PACU
* In the PACU, patients will have their pain assessed by the non-verbal FLACC pain scale, Figure 4.
* Pain scores will be recorded at 5, 30, 60, and 90 minutes' post-procedure as well as at the time of discharge from the PACU to home. These scores will be given by the PACU nursing staff and separately by the parents for consistency in scoring the post-operative period of the patient.
* The nursing staff will be given an in-service education about the trial and using the FLACC scoring scale. They will also be given the opportunity to score patients alongside a provider during the initial pilot of the study with either the pediatric urologist, pediatric urology fellow, or pediatric anesthesiologist. We will also be collaborating with a member of the PACU staff to serve as part of the research personnel (potentially a nurse who has an academic interest or seeking an opportunity to further their education in research) to further offer consistency of PACU nursing staff education and transition of information to the patients' parents. This will hopefully decrease the concern for inconsistency of parent education and nursing PACU scoring of patient's pain.
* In addition, the amount of narcotic pain medication required (if any) will be documented. Any requirement for narcotic pain medication in PACU will be considered a failure of the block and these patients will be assigned a pain score of zero out of 10 on the FLACC scale.
* We will also monitor patients for emergence delirium and if the patient required a bolus of propofol or dexmedetomidine in the PACU. This will be reported in the medical record and factored in when interoperating results.
* The patient will be discharged from PACU with a prescription for the weight-based dosage of acetaminophen and ibuprofen. This will allow the medications to be given at the appropriate weight dosage and for the patients to potentially have the agents covered by the insurance or bought over the counter.
* Patients will also be given a prescription for oxybutynin to use for bladder spasm (catheter associated pain) that will be weight based to use on a PRN basis.

  3. Post-Operative Scoring using the FLACC non-verbal pain scale
* The parents will be asked to assess their child's pain using the FLACC scale in 6 hour intervals (while awake and if sleeping will be assigned a 0 for that time period). If the child has a score of >4 the patient will be given a weight calculated dose of acetaminophen or ibuprofen alternating each time a score > 4 occurs. If the patient is experiencing a score >7 then patient will be administered a weight based dosage of oral narcotic medication. [20]
* All patients will be sent home with PRN oral acetaminophen and Ibuprofen pain medication per our department's standard practice. PACU RNs will be blinded to the block that each patient will receive. The anesthesiologist and urologist will be the only people who are aware of the randomization for patient safety concerns, but will never be assigning a patient FLACC score therefore this should not impact results.
* The caregiver of the child will be given a copy of the FLACC and asked to record their child's score in 6 hour intervals and any PRN pain medications administered and the score at the time of medication administration.
* The highest score given in the first 24, 48, 72 hours will be used as the values for analysis for Time 1, 2, and 3 respectively. We will also look at the total sum of pain scores per 24-hour period. (If the parents give more than 1 score in a 6-hour window then the highest score from that period will be used in the calculation).
* During the randomization process, there will be random patients (most likely every 4th patient for a total of 25 patients throughout the course of the trial) selected for an additional post-operative phone call at 24 hours. This phone call will be done by a member of the research team via FaceTime or Skype, where the ability to visualize the patient and award a FLACC score alongside the parent/caregiver can be conducted. This will hopefully be able to support the concept of parents being educated in the scoring system in hopes of eliminating intraoperative scoring error between families when compared to the research team member.
* Each family will receive a standard phone call at 72 hours to verify any adverse events, presentations to ER or another provider prior to scheduled follow up appointment, requirements for pain medication, and to collect the parentally recorded pain scale data at their follow up appointment which occurs at 1 week (5-10 days postoperatively) when the patient presents for catheter removal. At that time, the parents will be interviewed and asked about the postoperative course and any complications such as UTI, fever, or adverse events as defined above.
* The parents will be given a survey after the initial post-operative course to inquire about their experience and their opinion on their child's post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 6 months to 24 months of all races and ethnicities that have hypospadias requiring surgical intervention and post-operative urethral catheterization.

Exclusion Criteria:

* Males who are not age 6 mo. to 24 months, those who do not have a diagnosis of hypospadias, those who have an ASA class of 3 or greater or known liver or renal impairment, or who have an allergy to local anesthetics such as lidocaine, bupivacaine, etc.

Ages: 6 Months to 24 Months | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Difference in Mean Pain Scores recorded over the first 72 hours following surgery between the 2 arms | For 72 hours following surgery
  Pain levels as indicated by the non-verbal Face, Legs, Activity, Cry, Consolability (FLACC) pain scale with liposomal vs standard bupivacaine. The scale allots each area mentioned in the acronym 0-2 points for a total scale of 0-10. 0 indicates no pain with greater scores indicating higher pain severity.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Peters, MD, Principal Investigator — UT Southwestern

IPD SHARING:
Plan to Share IPD: Yes
An adequate plan is in place to protect the patient identifiers. The plan includes that the electronic datasheet will reside in the researchers UTSW secure O:drive and will not be transmitted outside the institution as this is a PI-initiated trial. The UTSW HRPP/IRB offices, Children's and UTSW offices of research administration, and any state or federal monitors may be given access to study records or data on site, as necessary. The data will be password protected, passwords will be changed on a regular basis, access to the data will be restricted to the research team only, and all paper records will be kept in locked file cabinets and access limited to authorized personnel only. The identifiers will be destroyed after the de-identified results have been submitted for publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Until trial completion and data publication in 2023
Access Criteria: Research team only

REFERENCES:
- [Background] Dadure, C., et al., Regional Anesthesia in Children in Miller's Anesthesia, R.E. Miller, Lars. Fleisher,Lee. Wiener-Kronish,Jeanine. Cohen,Neal. Young,William., Editor. 2015, Elsevier: Philadelphia, PA. p. 2706-2756
- [Background] Tutuncu AC, Kendigelen P, Ashyyeralyeva G, Altintas F, Emre S, Ozcan R, Kaya G. Pudendal Nerve Block Versus Penile Nerve Block in Children Undergoing Circumcision. Urol J. 2018 May 3;15(3):109-115. doi: 10.22037/uj.v0i0.4292. PMID 29299888
- [Background] Naja Z, Al-Tannir MA, Faysal W, Daoud N, Ziade F, El-Rajab M. A comparison of pudendal block vs dorsal penile nerve block for circumcision in children: a randomised controlled trial. Anaesthesia. 2011 Sep;66(9):802-7. doi: 10.1111/j.1365-2044.2011.06753.x. Epub 2011 Jul 25. PMID 21790518
- [Background] Gray, H., Anatomy of the human body. 20 ed. 1918, Philidelphia: Lea & Febiger. 968
- [Background] Richard BM, Ott LR, Haan D, Brubaker AN, Cole PI, Nelson KG, Ross PE, Rebelatto MC, Newton PE. The safety and tolerability evaluation of DepoFoam bupivacaine (bupivacaine extended-release liposome injection) administered by incision wound infiltration in rabbits and dogs. Expert Opin Investig Drugs. 2011 Oct;20(10):1327-41. doi: 10.1517/13543784.2011.611499. Epub 2011 Aug 26. PMID 21867476
- [Background] Chahar P, Cummings KC 3rd. Liposomal bupivacaine: a review of a new bupivacaine formulation. J Pain Res. 2012;5:257-64. doi: 10.2147/JPR.S27894. Epub 2012 Aug 14. PMID 23049275
- [Background] Mantripragada S. A lipid based depot (DepoFoam technology) for sustained release drug delivery. Prog Lipid Res. 2002 Sep;41(5):392-406. doi: 10.1016/s0163-7827(02)00004-8. PMID 12121719
- [Background] Mowat JJ, Mok MJ, MacLeod BA, Madden TD. Liposomal bupivacaine. Extended duration nerve blockade using large unilamellar vesicles that exhibit a proton gradient. Anesthesiology. 1996 Sep;85(3):635-43. doi: 10.1097/00000542-199609000-00024. PMID 8853095
- [Background] Ostro MJ, Cullis PR. Use of liposomes as injectable-drug delivery systems. Am J Hosp Pharm. 1989 Aug;46(8):1576-87. PMID 2672806
- [Background] Dullenkopf A, Borgeat A. [Local anesthetics. Differences and similarities in the "-cains"]. Anaesthesist. 2003 Apr;52(4):329-40. doi: 10.1007/s00101-003-0463-5. German. PMID 12715136
- [Background] Pacira Pharmaceuticals. Exparel: Bupivacaine Liposome Injectable Suspension. [Prescribing Information]. Parsippany, NJ [Accessed August 23, 2018]. Available from: https://www.exparel.com/hcp/prescriptioninformation.pdf.
- [Background] Wolfe JW, Butterworth JF. Local anesthetic systemic toxicity: update on mechanisms and treatment. Curr Opin Anaesthesiol. 2011 Oct;24(5):561-6. doi: 10.1097/ACO.0b013e32834a9394. PMID 21841477
- [Background] Bergese SD, Onel E, Morren M, Morganroth J. Bupivacaine extended-release liposome injection exhibits a favorable cardiac safety profile. Reg Anesth Pain Med. 2012 Mar-Apr;37(2):145-51. doi: 10.1097/AAP.0b013e31823d0a80. PMID 22266897
- [Background] Golf M, Daniels SE, Onel E. A phase 3, randomized, placebo-controlled trial of DepoFoam(R) bupivacaine (extended-release bupivacaine local analgesic) in bunionectomy. Adv Ther. 2011 Sep;28(9):776-88. doi: 10.1007/s12325-011-0052-y. Epub 2011 Aug 12. PMID 21842428
- [Background] Bramlett K, Onel E, Viscusi ER, Jones K. A randomized, double-blind, dose-ranging study comparing wound infiltration of DepoFoam bupivacaine, an extended-release liposomal bupivacaine, to bupivacaine HCl for postsurgical analgesia in total knee arthroplasty. Knee. 2012 Oct;19(5):530-6. doi: 10.1016/j.knee.2011.12.004. Epub 2012 Jan 28. PMID 22285545
- [Background] Davidson EM, Barenholz Y, Cohen R, Haroutiunian S, Kagan L, Ginosar Y. High-dose bupivacaine remotely loaded into multivesicular liposomes demonstrates slow drug release without systemic toxic plasma concentrations after subcutaneous administration in humans. Anesth Analg. 2010 Apr 1;110(4):1018-23. doi: 10.1213/ANE.0b013e3181d26d2a. PMID 20357145
- [Background] Gorfine SR, Onel E, Patou G, Krivokapic ZV. Bupivacaine extended-release liposome injection for prolonged postsurgical analgesia in patients undergoing hemorrhoidectomy: a multicenter, randomized, double-blind, placebo-controlled trial. Dis Colon Rectum. 2011 Dec;54(12):1552-9. doi: 10.1097/DCR.0b013e318232d4c1. PMID 22067185
- [Background] Smoot JD, Bergese SD, Onel E, Williams HT, Hedden W. The efficacy and safety of DepoFoam bupivacaine in patients undergoing bilateral, cosmetic, submuscular augmentation mammaplasty: a randomized, double-blind, active-control study. Aesthet Surg J. 2012 Jan;32(1):69-76. doi: 10.1177/1090820X11430831. Epub 2011 Dec 16. PMID 22179931
- [Background] Day KM, Nair NM, Sargent LA. Extended Release Liposomal Bupivacaine Injection (Exparel) for Early Postoperative Pain Control Following Palatoplasty. J Craniofac Surg. 2018 Jul;29(5):e525-e528. doi: 10.1097/SCS.0000000000004591. PMID 29762332
- [Background] Manworren RC, Hynan LS. Clinical validation of FLACC: preverbal patient pain scale. Pediatr Nurs. 2003 Mar-Apr;29(2):140-6. PMID 12723828